CLINICAL TRIAL: NCT05387005
Title: Identification of the Optimal Screening Strategy for Gastric Cancer Prevention
Brief Title: Screening Strategy for Gastric Cancer Prevention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 202203064RINC
Record Dates: First submitted 2022-04-28; First posted 2022-05-24 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: H. Pylori Infection
Keywords: H. pylori; screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- UBT (Experimental)
  Interventions: Diagnostic Test: UBT
- HpSA (Experimental)
  Interventions: Diagnostic Test: HPSA
- Standard method (Experimental)
  Interventions: Diagnostic Test: UBT and HPSA
- Two-stage screening method (Experimental)
  Interventions: Diagnostic Test: Serology (two stage)

INTERVENTIONS:
Diagnostic Test: UBT — H. pylori diagnostic test: C13 urea breath test
  Arms: UBT
Diagnostic Test: HPSA — H. pylori diagnostic test: H. pylori stool antigen test
  Arms: HpSA
Diagnostic Test: UBT and HPSA — H. pylori diagnostic tests: H. pylori serology test, C13 urea breath test
  Arms: Standard method
Diagnostic Test: Serology (two stage) — H. pylori diagnostic test: If H. pylori serology is positive, confirmation UBT will be done.
  Arms: Two-stage screening method

SUMMARY:
There are still some unsolved questions regarding population-based screening program for H. pylori infection to prevent gastric cancer, such as how to perform the optimal screening strategies. A prospective, randomized trial will be conducted to compare the acceptability, compliance (/adherence), and accuracy of diagnostic tests in a population-based H. pylori screening and gastric cancer prevention program.

Initially, we planned to recruit 10,000 adults aged ≥20 years who had not previously undergone H. pylori screening or treatment. Eligible participants were to be randomly allocated in a 1:1:1:1 ratio to one of four groups, each receiving a different combination of diagnostic tests. However, a preliminary analysis led to a recalculation of the required sample size. Following the approval of an Institutional Review Board (IRB) amendment, enrollment was discontinued for Group B (HpSA method) and Group D (Two-stage screening method). The final number of participants enrolled in Group B and Group D was 852 and 851, respectively. Groups A (UBT method) and Group C (standard method) will continue to enroll participants through an additional 1:1 randomization until each group reaches a total of 1,350 participants.

DETAILED DESCRIPTION:
Background: There are still some unsolved questions regarding population-based screening program for H. pylori infection to prevent gastric cancer, such as how to perform the optimal screening strategies.

Objective: A prospective, randomized trial will be conducted to compare the acceptability, compliance (/adherence), and accuracy of C13 UBT and HpSA in a population-based H. pylori screening and gastric cancer prevention program.

Methods：Open labeled, randomized controlled trial Initially, the investigators will recruit adults with age of ≥20 years who have not received H. pylori screening or treatment. Eligible patients were randomly 1:1:1:1 allocated to (A) The carbon-13 urea breath test (C13 UBT), (B) H. pylori stool antigen test (Vstrip® HpSA), (C) Standard method (Both C13 UBT and HpSA), (D) Two-stage screening method (serology screening only, and then C13 UBT for confirmation if serology test is positive). However, a preliminary analysis led to a recalculation of the required sample size. Following the approval of an Institutional Review Board (IRB) amendment, enrollment was discontinued for Group B and Group D. The final number of participants enrolled in Group B and Group D was 852 and 851, respectively. Groups A and Group C will continue to enroll participants through an additional 1:1 randomization until each group reaches a total of 1,350 participants.

Outcome analysis:

1. Detection rate of H. pylori infection
2. To compare the compliance(/adherence) of screening tests for H. pylori infection in the two randomized groups.
3. To assess the diagnostic accuracy of these tests.
4. To verify the compliance(/adherence) and feasibility of this two-stage screening method
5. Long-term Outcomes: To assess the risk reduction of gastric cancer

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20 years or older
* Never screened and treated for H. pylori infection

Exclusion Criteria:

* Ever undergone gastrectomy
* Patients with gastric cancer
* Have been screened or tested for H. pylori infection
* Ever received H. pylori eradication therapy
* Have taken proton pump inhibitor within two weeks
* Have taken antibiotics within two weeks

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4403 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Detection rates of H. pylori infection | 2-8 weeks
  The positivity rate of H. pylori infection between different study arms, respectively in ITT and PP analysis.

SECONDARY OUTCOMES:
The compliance(/adherence) of screening tests for H. pylori infection in the two randomized groups | 2 weeks to 1 year
  Completion rates of the study (from enrollment to the diagnosis of H. pylori; from enrollment to the treatment of H. pylori infection.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No